CLINICAL TRIAL: NCT03151772
Title: Drug Level and Investigation of Novel Substances Indicated Downstream Effect in Glioblastoma
Brief Title: Bioavailability of Disulfiram and Metformin in Glioblastomas
Acronym: INSIDE
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Problems with including patients
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Asgeir S. Jakola, Associate professor, neurosurgeon, Sahlgrenska University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1144-16
Record Dates: First submitted 2017-05-09; First posted 2017-05-12 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Disulfiram; Metformin

STUDY DESIGN:
Intervention Model Description: Bioavailability study with an adaptive design (evaluation after 5 patients up to a total maximum of 20 patients in each arm). Experimental therapy not to be combined and not any comparison between therapies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Disulfiram (Experimental): Disulfiram 200 mg twice daily and copper 2,5 mg once daily. For bioavailability purpose only, treatment is withdrawn postoperatively
  Interventions: Drug: Disulfiram
- Metformin (Experimental): Metformin 850 mg x 3 daily. For bioavailability purpose only, treatment is withdrawn postoperatively
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Disulfiram — 200 mg disulfiram two times daily and 2,5 mg copper once daily taken preoperatively
  Arms: Disulfiram
Drug: Metformin — Metformin 850 mg x 3 taken preoperatively
  Arms: Metformin

SUMMARY:
Neuro-oncological trials may fail due to the drug never getting to the intended target (i.e. within the tumor micro environment). Also, changes' occurring in tumor cells when removed from patients and grown in-vitro is another limiting factor influencing the clinical success.

Important questions are therefore:

1. Does the drug get there?
2. Does the drug do what it is intended to do?

To improve chances of clinical success there is a need for rational and intelligent selection of potential drugs in future trials. This is an initiative for analyzing tumor concentration of preoperative administered repurposed drugs

ELIGIBILITY:
Inclusion Criteria:

The subjects must fulfill all the following inclusion criteria to be eligible for participation in the study, unless otherwise specified:

1. A suspected glioblastoma (based on MRI) or recurrent glioblastoma undergoing surgical resection.
2. Elective surgical indication
3. Age 18 years or older.
4. Karnofsky performance status of 60 - 100 (see attachment 3).
5. Not receiving another experimental treatment for glioblastoma at the moment of inclusion.
6. Able to take oral medications.
7. No known allergy to substance
8. Absolute neutrophil count ≥ 1,500/mcL and platelets ≥ 100,000/mcL

Exclusion Criteria:

General

1. Other likely diagnosis than glioblastoma based on MRI.
2. Pregnant and/or breastfeeding.
3. Women of childbearing potential who do not have a negative pregnancy test (not older than 14 days) before inclusion.
4. History of active liver disease, including chronic active hepatitis, viral hepatitis (hepatitis B, C and CMV), cholestatic jaundice of any etiology or toxic hepatitis or inadequate hepatic function, defined as baseline ASAT and ALAT > 1.5 X upper institutional limit and/or bilirubin > 1.5 X upper institutional limit.
5. Suspected significant raised intracranial pressure or other indication for emergent surgery
6. Unfit for participation for any other reason judged by the including physician.

Specific additional exclusions criteria for disulfiram

1. History of uncontrolled hypertension (i.e. systolic BP > 180 mmHg) and a diagnosis of congestive heart failure
2. History of psychiatric conditions (e.g. depression, psychosis, schizophrenia) or dementia.
3. History of Wilson's disease or family member with Wilson's disease (unless excluded as a carrier by genetic test).
4. History of hemochromatosis or family member with hemochromatosis (unless excluded as a carrier by genetic test).
5. Nickel hypersensitivity (disulfiram mobilize nickel causing a brief increase in nickel concentrations before excretion. The initial increase may lead to hepatitis and predisposed patients).7
6. Need for metronidazole, warfarin and/or theophylline medication (the metabolism may be influenced by disulfiram).
7. Patients who are taking medications metabolized by cytochrome P450 2E1, including chlorzoxazone or halothane and its derivatives (phenytoin, phenobarbital, chlordiazepoxide, imipramine, diazepam, isoniazid, metronidazole, warfarin, amitriptyline within 14 days prior to the first dose of disulfiram. Of note, lorazepam and oxazepam are not affected by the P450 system and are not contraindicated with disulfiram).
8. Addiction to alcohol or drugs. Alcohol must be avoided.
9. Serum/plasma copper and serum ceruloplasmin outside institutional limits. a. However increased levels are seen together with ongoing acute phase reaction as determined by elevated C-reactive protein (ceruloplasmin is elevated as part of the same process) it is possible to retest after normalization of C-reactive protein.

Specific additional exclusions criteria for metformin

1. Diabetic patients or other patients where treating physician and/or anesthesiologist consider may have an increased risk for lactic acidosis per- and postoperatively
2. Known renal failure, renal risk factors (including single kidney, donor kidney, polycystic kidneys) or estimated glomerular filtration rate below 80 ml/min.
3. Congestive heart failure
4. Scheduled diagnostic work-up where contrast medium containing iodine is indicated
5. Concomitant use of NSAIDs (risk of renal injury)
6. Risk of dehydration judged by the treating physician (e.g. when symptoms include vomiting)
7. Alcohol must be avoidance during treatment (increased risk of lactic acidosis)
8. Treatment with diuretics as they may increase risk of lactic acidosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-09-24 (Actual)

PRIMARY OUTCOMES:
Bioavailabilty disulfiram | At time of surgery
  Concentration of disulifram-copper complex available in glioblastoma compared to blood
Bioavailabilty of metformin | At time of surgery
  Concentration of metformin available in glioblastoma compared to blood

CONTACTS AND LOCATIONS:
Overall Officials: Asgeir S Jakola, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No